CLINICAL TRIAL: NCT00072462
Title: International Breast Cancer Intervention Study II (IBIS-II) (DCIS)
Brief Title: Adjuvant Tamoxifen Compared With Anastrozole in Treating Postmenopausal Women With Ductal Carcinoma In Situ
Acronym: IBIS-II DCIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISRCTN37546358; EU-20226; BIG-5-02; IBCSG-31-03-DCIS; ISRCTN31488319
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
Keywords: ductal breast carcinoma in situ; breast cancer in situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ | interventions — Tamoxifen; Anastrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anastrozole (Active Comparator)
  Interventions: Drug: Anastrozole
- Tamoxifen (Active Comparator)
  Interventions: Drug: tamoxifen citrate

INTERVENTIONS:
Drug: tamoxifen citrate — Tamoxifen 20mg + Anastrozole placebo
  Other Names: Nolvadex
  Arms: Tamoxifen
Drug: Anastrozole — Anastrozole 1mg + Tamoxifen placebo
  Other Names: Arimidex
  Arms: Anastrozole

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using either tamoxifen or anastrozole may fight breast cancer by blocking the use of estrogen. It is not yet known whether tamoxifen is more effective than anastrozole in preventing breast cancer after surgery for ductal carcinoma in situ.

PURPOSE: This randomized phase III trial is studying how well adjuvant tamoxifen works compared to anastrozole in treating postmenopausal women who have undergone surgery to remove ductal carcinoma in situ.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of adjuvant tamoxifen vs anastrozole, in terms of local control and prevention of contralateral disease, in postmenopausal women with locally excised ductal carcinoma in situ.
* Compare side effect profiles of these drugs in these patients.

Secondary

* Compare the efficacy of these drugs, according to the receptor status of the primary or recurrent cancer in these patients.
* Compare the rate of breast cancer recurrence and growth of new contralateral tumors after cessation of treatment with these drugs in these patients.
* Compare breast cancer mortality in patients treated with these drugs.
* Compare the effect of these drugs on other cancers, cardiovascular disease, fracture rates, and non-breast cancer deaths in these patients.
* Compare the tolerability and acceptability of side effects experienced by patients treated with these drugs.

OUTLINE: This is a randomized, double-blind, multicentre study. Patients are stratified according to participating centre. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral tamoxifen and oral placebo once daily.
* Arm II: Patients receive oral anastrozole and oral placebo once daily. In both arms, treatment continues for 5 years in the absence of disease recurrence or unacceptable toxicity.

Patients are followed annually for 5 years and a further 5 years (minimum) off treatment.

Peer Reviewed and Funded by Cancer Research UK. Sponsored by Queen Mary University of London

ACTUAL ACCRUAL: A total of 2,980 patients were accrued for this study over 9 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of ductal carcinoma in situ within the past 6 months

  * Locally excised with tumor-free margins at least 1 mm
* Hormone receptor status:

  * Estrogen or progesterone receptor positive

    * Equal to or greater than 5% positive cells

PATIENT CHARACTERISTICS:

Age

* 40 to 70

Sex

* Female

Menopausal status

* Postmenopausal, defined as meeting at least 1 of the following criteria:

  * Over age 60
  * Prior bilateral oophorectomy
  * Age 60 or under with a uterus AND amenorrhea for at least the past 12 months
  * Age 60 or under without a uterus AND follicle-stimulating hormone greater than 20 IU/L

Performance status

* Not specified

Life expectancy

* At least 10 years

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Cardiovascular

* No prior deep vein thrombosis
* No prior transient ischemic attack
* No prior cerebrovascular accident

Pulmonary

* No prior pulmonary embolism

Other

* No unexplained postmenopausal bleeding
* No other cancer within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No other concurrent medical condition that would preclude study therapy, place the patient at unusual risk, or confound study results
* No evidence of osteoporosis
* Fragility fractures within the spine allowed if T-score level is greater than -4 and consist of no more than 2 fractures
* Psychologically and physically suitable for 5 years of study therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* No prior or concurrent tamoxifen use lasting more than 6 months unless treatment was completed more than 5 years ago. Women in IBIS-I can join if off trial therapy for at least 5 years.
* No prior or concurrent raloxifene use lasting more than 6 months unless treatment was completed more than 5 years ago.
* No other prior or concurrent selective estrogen-receptor modulator use lasting more than 6 months unless treatment was completed more than 5 years ago
* No concurrent systemic estrogen-based hormone replacement therapy, including vaginal estrogen preparations

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics
* No prior mastectomy
* No planned prophylactic mastectomy

Other

* At least 3 months since prior unapproved or experimental agents
* No concurrent anticoagulants

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2980 (Actual)
Dates: Start 2003-09; Primary Completion 2015-12 (Actual); Study Completion 2021-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack Cuzick, PhD, Study Chair — Queen Mary University of London; Anthony Howell, Study Chair — University of Manchester
Locations (97):
- Australia, Newcastle, Australia
- Austrian Breast & Colorectal Cancer Study Group, Vienna, Austria
- Belgium, Leuven, Belgium
- Chile, Santiago, Chile
- France (20):
  - Institut Sainte Catherine, Avignon
  - Institut Bergonie, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Clinique Tivoli, Bordeaux
  - CHU Hopital A. Morvan, Brest
  - Centre Regional Francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon
  - Centre Hospitalier de Lagny, Lagny-sur-Marne
  - CMC Les Ormeaux, Le Havre
  - Centre Oscar Lambret, Lille
  - Centre Hospital Regional Universitaire de Limoges, Limoges
  - Centre Hospitalier de Mulhouse, Mulhouse
  - Centre Regional Rene Gauducheau, Nantes
  - Clinique Saint - Pierre, Perpignan
  - Institut Jean Godinot, Reims
  - Centre Eugene Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany, Neu-Isenburg, Germany
- Hungary, Szeged, Hungary
- Ireland (8):
  - Cork Infirmary, Cork
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - St. Vincent's University Hospital, Dublin
  - University College Hospital, Galway
  - Mid-Western Regional Hospital, Limerick
  - Sligo General Hospital, Sligo
  - The Adelaide and Meath Hospital, Tallaght
- European Institute of Oncology, Milan, Italy
- Sir Paul Boffa Hospital,, Floriana, Malta
- Sweden, Lund, Sweden
- Switzerland (9):
  - Inselspital Bern, Bern
  - Oncocare Sonnenhof-Klinik Engeriedspital, Bern
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonspital, Lucerne
  - Ospedale Beata Vergine, Mendrisio
  - Tumor Zentrum ZeTup St. Gallen und Chur, Sankt Gallen
  - Switzerland(St. Gallen), Sankt Gallen
  - Regionalspital, Thun
- Turkey(Istanbul University), Istanbul, Turkey (Türkiye)
- United Kingdom (50):
  - Frenchay Hospital, Bristol, England
  - Colchester General Hospital, Colchester, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Royal Liverpool University Hospital, Liverpool, England
  - Whittington Hospital, London, England
  - St. Thomas' Hospital, London, England
  - Christie Hospital, Manchester, England
  - Newcastle Upon Tyne Hospitals NHS Trust, Newcastle upon Tyne, England
  - Nottingham City Hospital, Nottingham, England
  - Royal South Hants Hospital, Southampton, England
  - Centre for Cancer Research and Cell Biology at Queen's University Belfast, Belfast, Northern Ireland
  - St. Bartholomew's Hospital, London, Please Select
  - Royal Marsden Hospital, London, Please Select
  - Ninewells Hospital, Dundee, Scotland
  - Royal Infirmary of Edinburgh at Little France, Edinburgh, Scotland
  - University Hospital of Wales, Cardiff, Wales
  - Aberdeen Royal Infirmary, Aberdeen
  - Tameside General Hospital, Ashton-under-Lyne
  - Royal Bolton Hospital, Bolton
  - Royal Bournemouth Hospital, Bournemouth
  - St Lukes Hospital, Bradford
  - Royal Sussex County Hospital, Brighton
  - Bristol Infirmary, Bristol
  - Queens Hospital Burton, Burton
  - Cheltenham General Hospital, Cheltenham
  - Countess of Chester Hospital, Chester
  - Derbyshire Royal Infirmary, Derby
  - St Margaret's Hospital, Epping
  - Royal Devon and Exeter Hospital, Exeter
  - Frimley Park Hospital NHS Trust, Frimley
  - Grantham & District Hospital, Grantham
  - Conquest Hospital, The Ridge, Hastings
  - Huddersfield Royal Infirmary, Huddersfield
  - Castle Hill Hospital, Hull
  - Airedale General Hospital, Keighley
  - Leeds St James., Leeds
  - Lincoln County Hospital, Lincoln
  - Derriford Hospital, Plymouth
  - Royal Hospital Haslar, Portsmouth
  - Scarborough NHS Trust, Scarborough
  - Weston Park Hospital, Sheffield
  - Staffordshire General Hospital, Stafford
  - Singleton Hospital, Swansea
  - Treliske Royal Cornwall Hospital, Truro
  - Clayton Hospital, Northgate, Wakefield
  - Welwyn Garden City Hospital, Welwyn
  - Wishaw General Hospital, Wishaw
  - Worthing Hospital, Worthing
  - Yeovil District Hospital, Yeovil
  - York Hospital, York

REFERENCES:
- [Background] Juraskova I, Butow P, Lopez A, Seccombe M, Coates A, Boyle F, McCarthy N, Reaby L, Forbes JF. Improving informed consent: pilot of a decision aid for women invited to participate in a breast cancer prevention trial (IBIS-II DCIS). Health Expect. 2008 Sep;11(3):252-62. doi: 10.1111/j.1369-7625.2008.00498.x. PMID 18816321
- [Background] Forbes JF, Sestak I, Howell A, Bonanni B, Bundred N, Levy C, von Minckwitz G, Eiermann W, Neven P, Stierer M, Holcombe C, Coleman RE, Jones L, Ellis I, Cuzick J; IBIS-II investigators. Anastrozole versus tamoxifen for the prevention of locoregional and contralateral breast cancer in postmenopausal women with locally excised ductal carcinoma in situ (IBIS-II DCIS): a double-blind, randomised controlled trial. Lancet. 2016 Feb 27;387(10021):866-73. doi: 10.1016/S0140-6736(15)01129-0. Epub 2015 Dec 11. PMID 26686313
- [Background] Sestak I, Smith SG, Howell A, Forbes JF, Cuzick J. Early participant-reported symptoms as predictors of adherence to anastrozole in the International Breast Cancer Intervention Studies II. Ann Oncol. 2018 Feb 1;29(2):504-509. doi: 10.1093/annonc/mdx713. PMID 29126161
- See also: Clinical trial summary from Cancer Research UK Website — http://www.cancerresearchuk.org/about-cancer/find-a-clinical-trial/a-trial-looking-at-tamoxifen-or-anastrozole-in-postmenopausal-women-with-ductal-carcinoma-in-situ-of-the-breast
- See also: IBIS-II website — https://www.ibis-trials.org/thetrials/ibistrials/ibis-2-dcis

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anastrozole | Tamoxifen
Started | 1471 | 1509
Completed | 1449 | 1489
Not Completed | 22 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anastrozole | Tamoxifen | Total
Number analyzed (Participants) | 1471 | 1509 | 2980
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1139 | 1171 | 2310
  >=65 years | 332 | 338 | 670
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60.4 [56.4 to 64.7] | 60.3 [55.8 to 64.5] | 60.3 [56.1 to 64.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1471 | 1509 | 2980
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 4 | 4 | 8
  United Kingdom | 429 | 460 | 889
  Italy | 165 | 158 | 323
  Australia | 76 | 92 | 168
  Switzerland | 19 | 26 | 45
  Belgium | 54 | 50 | 104
  Chile | 9 | 8 | 17
  Finland | 4 | 3 | 7
  Ireland | 42 | 36 | 78
  France | 211 | 215 | 426
  Germany | 386 | 393 | 779
  Hungary | 7 | 8 | 15
  Malta | 2 | 2 | 4
  New Zealand | 4 | 6 | 10
  Turkey | 7 | 8 | 15
  Austria | 51 | 39 | 90
  India | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Breast Cancer Recurrence, Including Recurrent DCIS and New Contralateral Tumours
Time Frame: Date of the breast cancer occurrence is defined as the date of the confirmation of the specific event (from randomisation to date of occurrence). Data presented is from randomisation to study completion, median follow-up was 11.6 years (IQR: 9.9-13.5).
Measure: Count of Participants; unit: Participants
Arm/Group | Anastrozole | Tamoxifen
Number analyzed (Participants) | 1449 | 1489
Participants | 103 | 120
Statistical Analysis 1: Comparison: Anastrozole vs Tamoxifen; Test type: Superiority; p = 0.33, Regression, Cox; Univariate; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.67 to 1.14], Standard Deviation 0.12
Statistical Analysis 2: Comparison: Anastrozole vs Tamoxifen; Test type: Superiority; p = 0.33, Regression, Cox; Covariates included in model: Hormone Replacement Therapy use, Age, BMI, Use of radiotherapy, Extent of margins, Grade(categorical: low, medium, high); Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.66 to 1.15], Standard Deviation 0.12

2. Secondary Outcome: Number of Participants With ER+ Breast Cancer Recurrence, Including Recurrent DCIS and New Contralateral Tumours
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Anastrozole | Tamoxifen
Number analyzed (Participants) | 1449 | 1489
Participants | 58 | 82
Statistical Analysis 1: Comparison: Anastrozole vs Tamoxifen; Test type: Superiority; p = 0.06, Regression, Cox; Univariate; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.52 to 1.01], Standard Deviation 0.12
Statistical Analysis 2: Comparison: Anastrozole vs Tamoxifen; Test type: Superiority; p = 0.09, Regression, Cox; [statistical method as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.52 to 1.05], Standard Deviation 0.13

3. Secondary Outcome: Number of Participants With ER- Breast Cancer Recurrence
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Anastrozole | Tamoxifen
Number analyzed (Participants) | 1449 | 1489
Participants | 24 | 15
Statistical Analysis 1: Comparison: Anastrozole vs Tamoxifen; Test type: Superiority; p = 0.13, Regression, Cox; Univariate; Hazard Ratio (HR) = 1.64, 95% CI 2-sided [0.75 to 2.84], Standard Deviation 0.54
Statistical Analysis 2: Comparison: Anastrozole vs Tamoxifen; Test type: Superiority; p = 0.26, Regression, Cox; [statistical method as in outcome 1, analysis 2]; Hazard Ratio (HR) = 1.46, 95% CI 2-sided [0.75 to 2.84], Standard Deviation 0.50

4. Secondary Outcome: Number of Breast Cancer Deaths
Time Frame: Date of the death is defined as the date of the confirmation of the specific event (from randomisation to date of occurrence). Data presented is from randomisation to study completion, median follow-up was 11.6 years (IQR: 9.9-13.5).
Measure: Count of Participants; unit: Participants
Arm/Group | Anastrozole | Tamoxifen
Number analyzed (Participants) | 1449 | 1489
Participants | 3 | 3
Statistical Analysis 1: Comparison: Anastrozole vs Tamoxifen; Test type: Superiority; p = 0.97, Regression, Cox; Univariate; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.21 to 5.11]
Statistical Analysis 2: Comparison: Anastrozole vs Tamoxifen; Test type: Superiority; p = 0.93, Regression, Cox; [statistical method as in outcome 1, analysis 2]; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.22 to 5.36], Standard Deviation 0.88

5. Secondary Outcome: Number of Non-breast Cancer Deaths
Time Frame: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Anastrozole | Tamoxifen
Number analyzed (Participants) | 1449 | 1489
Participants | 59 | 65
Statistical Analysis 1: Comparison: Anastrozole vs Tamoxifen; Test type: Superiority; p = 0.67, Regression, Cox; Univariate; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.65 to 1.32], Standard Deviation 0.17
Statistical Analysis 2: Comparison: Anastrozole vs Tamoxifen; Test type: Superiority; p = 0.38, Regression, Cox; [statistical method as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.59 to 1.22], Standard Deviation 0.16

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from randomisation to study completion, median follow-up was 11.6 years (IQR: 9.9-13.5).
Arm/Group | Anastrozole | Tamoxifen
All-Cause Mortality (participants affected / at risk) | 62/1449 | 69/1489
Serious Adverse Events (participants affected / at risk) | 333/1449 | 371/1489
Other Adverse Events (participants affected / at risk) | 1323/1449 | 1380/1489
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anastrozole (N=1449) | Tamoxifen (N=1489)
Aortic dissection (Vascular disorders) | 0 | 1
Arterial stenosis (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1
Infarction (Vascular disorders) | 0 | 1
Venous insufficiency (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Arterial thrombosis limb (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 5 | 14
Pelvic venous thrombosis (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 4
Thrombosis (Vascular disorders) | 2 | 5
Venous thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 2
Hot flush (Vascular disorders) | 2 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 4
Phlebitis (Vascular disorders) | 0 | 2
Varicose ulceration (Vascular disorders) | 0 | 1
Varicose vein (Vascular disorders) | 3 | 1
Bunion operation (Surgical and medical procedures) | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 2 | 5
Joint arthroplasty (Surgical and medical procedures) | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 3 | 2
Rotator cuff repair (Surgical and medical procedures) | 1 | 0
Mammoplasty (Surgical and medical procedures) | 1 | 1
Aortic valve replacement (Surgical and medical procedures) | 0 | 1
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 | 1
Mitral valve replacement (Surgical and medical procedures) | 1 | 0
Thyroid operation (Surgical and medical procedures) | 0 | 1
Thyroidectomy (Surgical and medical procedures) | 1 | 1
Eye operation (Surgical and medical procedures) | 0 | 1
Abdominal hernia repair (Surgical and medical procedures) | 1 | 0
Appendicectomy (Surgical and medical procedures) | 1 | 1
Colectomy (Surgical and medical procedures) | 0 | 1
Hernia repair (Surgical and medical procedures) | 1 | 1
Laparotomy (Surgical and medical procedures) | 0 | 1
Rectal prolapse repair (Surgical and medical procedures) | 0 | 1
Cholecystectomy (Surgical and medical procedures) | 1 | 0
Meningioma surgery (Surgical and medical procedures) | 0 | 1
Spinal laminectomy (Surgical and medical procedures) | 0 | 1
Spinal operation (Surgical and medical procedures) | 1 | 0
Hysterectomy (Surgical and medical procedures) | 1 | 1
Oophorectomy (Surgical and medical procedures) | 0 | 1
Oophorectomy bilateral (Surgical and medical procedures) | 0 | 1
Salpingo-oophorectomy bilateral (Surgical and medical procedures) | 0 | 2
Uterine dilation and curettage (Surgical and medical procedures) | 0 | 1
Uterine operation (Surgical and medical procedures) | 0 | 1
Uterine tumour excision (Surgical and medical procedures) | 0 | 1
Nephrectomy (Surgical and medical procedures) | 1 | 1
Removal of inert matter from skin or subcutaneous tissue (Surgical and medical procedures) | 0 | 1
Scar excision (Surgical and medical procedures) | 0 | 1
Skin graft (Surgical and medical procedures) | 0 | 1
Cancer surgery (Surgical and medical procedures) | 0 | 1
Debridement (Surgical and medical procedures) | 1 | 0
Elective surgery (Surgical and medical procedures) | 1 | 0
Lesion excision (Surgical and medical procedures) | 0 | 2
Malignant tumour excision (Surgical and medical procedures) | 0 | 2
Wound closure (Surgical and medical procedures) | 0 | 1
Coronary artery bypass (Surgical and medical procedures) | 1 | 0
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Paget's disease of the breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carcinoid tumour of the caecum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant palate neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Oral cavity cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Rectosigmoid cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haematological malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Focal nodular hyperplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Hairy cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pleural mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Meningeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Intraocular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 6
Uterine polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 8
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Fallopian tube cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 7
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 2
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Inflammatory myofibroblastic tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Sarcoma uterus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Allergy to arthropod bite (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 1
Cardiac death (General disorders) | 0 | 1
Death (General disorders) | 14 | 10
Asthenia (General disorders) | 1 | 0
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 2 | 6
Disease progression (General disorders) | 2 | 1
Fatigue (General disorders) | 0 | 2
Hernia (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 1 | 1
Pain (General disorders) | 0 | 1
Polyp (General disorders) | 0 | 1
Swelling (General disorders) | 0 | 1
Pelvic mass (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 0
Panic attack (Psychiatric disorders) | 0 | 1
Panic disorder (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 4 | 4
Hallucination (Psychiatric disorders) | 0 | 1
Drug abuse (Psychiatric disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Breast haematoma (Reproductive system and breast disorders) | 1 | 0
Breast necrosis (Reproductive system and breast disorders) | 0 | 2
Breast pain (Reproductive system and breast disorders) | 0 | 1
Cervical cyst (Reproductive system and breast disorders) | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0
Cervical polyp (Reproductive system and breast disorders) | 0 | 3
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 6
Metrorrhagia (Reproductive system and breast disorders) | 1 | 2
Ovarian atrophy (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 3
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 1
Cystocele (Reproductive system and breast disorders) | 2 | 4
Endometrial disorder (Reproductive system and breast disorders) | 0 | 1
Endometrial dysplasia (Reproductive system and breast disorders) | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 12
Endometrial hypertrophy (Reproductive system and breast disorders) | 0 | 5
Rectocele (Reproductive system and breast disorders) | 1 | 2
Uterine atrophy (Reproductive system and breast disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 15
Uterine prolapse (Reproductive system and breast disorders) | 1 | 3
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 3 | 3
Vaginal disorder (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 3 | 4
Vaginal polyp (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 10 | 11
Cartilage injury (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 | 4
Femur fracture (Injury, poisoning and procedural complications) | 3 | 2
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 3
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 2 | 2
Hand fracture (Injury, poisoning and procedural complications) | 2 | 1
Hip fracture (Injury, poisoning and procedural complications) | 4 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 4 | 3
Joint dislocation (Injury, poisoning and procedural complications) | 2 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 3 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 3 | 1
Patella fracture (Injury, poisoning and procedural complications) | 1 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 1
Radius fracture (Injury, poisoning and procedural complications) | 3 | 2
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 3
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 2 | 3
Wrist fracture (Injury, poisoning and procedural complications) | 4 | 4
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 1
Radiation fibrosis - lung (Injury, poisoning and procedural complications) | 0 | 1
Radiation necrosis (Injury, poisoning and procedural complications) | 0 | 1
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 6 | 2
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Ligament injury (Injury, poisoning and procedural complications) | 2 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 2
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 1
Traumatic anuria (Injury, poisoning and procedural complications) | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Multiple drug overdose (Injury, poisoning and procedural complications) | 1 | 0
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Post procedural pulmonary embolism (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Wound decomposition (Injury, poisoning and procedural complications) | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 1
Heart rate increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 1
Investigation (Investigations) | 0 | 1
Blood glucose fluctuation (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 0 | 1
Arthroscopy (Investigations) | 1 | 0
Intraocular pressure increased (Investigations) | 0 | 1
Body temperature increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Cystoscopy (Investigations) | 1 | 0
Hysteroscopy (Investigations) | 0 | 1
Smear cervix abnormal (Investigations) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 5 | 4
Atrial flutter (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Bundle branch block left (Cardiac disorders) | 0 | 1
Bundle branch block right (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 2
Extrasystoles (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 3
Aortic valve incompetence (Cardiac disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 3
Angina pectoris (Cardiac disorders) | 2 | 4
Angina unstable (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 2 | 3
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 4 | 6
Cardiac failure (Cardiac disorders) | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0
Arachnoiditis (Nervous system disorders) | 0 | 1
Encephalitis (Nervous system disorders) | 1 | 0
Brain stem stroke (Nervous system disorders) | 1 | 0
Carotid artery occlusion (Nervous system disorders) | 1 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 2
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 4 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 10 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 10 | 3
Trigeminal neuralgia (Nervous system disorders) | 1 | 0
Multiple sclerosis (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 2
Migraine (Nervous system disorders) | 1 | 0
Amnesia (Nervous system disorders) | 0 | 2
Dementia Alzheimer's type (Nervous system disorders) | 2 | 0
Hemiparesis (Nervous system disorders) | 0 | 1
Paresis (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 1 | 0
Diabetic hyperosmolar coma (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 2
Paraesthesia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 4 | 1
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 1
Motor neurone disease (Nervous system disorders) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 1
Diabetic neuropathy (Nervous system disorders) | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0
Nerve compression (Nervous system disorders) | 0 | 1
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Cataract (Eye disorders) | 5 | 2
Cataract cortical (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 0 | 1
Ocular hypertension (Eye disorders) | 1 | 0
Open angle glaucoma (Eye disorders) | 0 | 1
Optic ischaemic neuropathy (Eye disorders) | 0 | 1
Eye irritation (Eye disorders) | 0 | 1
Keratitis (Eye disorders) | 1 | 0
Macular hole (Eye disorders) | 0 | 2
Papilloedema (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 2
Retinal tear (Eye disorders) | 1 | 0
Retinal vein occlusion (Eye disorders) | 1 | 0
Blindness unilateral (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Deafness unilateral (Ear and labyrinth disorders) | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Enterocele (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 1
Colonic polyp (Gastrointestinal disorders) | 1 | 0
Gingival hypoplasia (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0
Pancreatic disorder (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 3
Colitis ischaemic (Gastrointestinal disorders) | 2 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrooesophagitis (Gastrointestinal disorders) | 1 | 0
Ileitis (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 4
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 2 | 4
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Volvulus of small bowel (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 2
Intestinal ulcer (Gastrointestinal disorders) | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Splenic artery aneurysm (Gastrointestinal disorders) | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 3
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Kidney enlargement (Renal and urinary disorders) | 1 | 0
Renal artery thrombosis (Renal and urinary disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 3
Renal impairment (Renal and urinary disorders) | 1 | 0
Urethral disorder (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Incontinence (Renal and urinary disorders) | 1 | 1
Mixed incontinence (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Stress urinary incontinence (Renal and urinary disorders) | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 4
Cholecystitis acute (Hepatobiliary disorders) | 3 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 3 | 1
Gallbladder polyp (Hepatobiliary disorders) | 0 | 2
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Hepatic cyst (Hepatobiliary disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 15 | 11
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 2
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 3
Lumbar spine flattening (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 3 | 1
Back disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Autoimmune thyroiditis (Endocrine disorders) | 0 | 1
Goitre (Endocrine disorders) | 3 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 0
Thyroiditis (Endocrine disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Diabetic foot (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Folate deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
Breast cellulitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 2 | 1
Escherichia infection (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 1 | 0
Pneumococcal sepsis (Infections and infestations) | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1
Abdominal infection (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Arthritis infective (Infections and infestations) | 0 | 1
Breast abscess (Infections and infestations) | 1 | 4
Bronchiectasis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 0
Bronchopneumonia (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 5 | 3
Endocarditis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Infection (Infections and infestations) | 0 | 1
Kidney infection (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Mastitis (Infections and infestations) | 3 | 1
Meningitis (Infections and infestations) | 1 | 0
Nail infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 5 | 10
Postoperative wound infection (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 1
Sialoadenitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 4 | 0
Urosepsis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 2
Herpes ophthalmic (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 2 | 0
Vestibular neuronitis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anastrozole (N=1449) | Tamoxifen (N=1489)
Ankle fracture (Injury, poisoning and procedural complications) | 9 | 10
Bone fragmentation (Injury, poisoning and procedural complications) | 1 | 0
Bursa injury (Injury, poisoning and procedural complications) | 0 | 1
Cartilage injury (Injury, poisoning and procedural complications) | 1 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 4
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 14 | 17
Forearm fracture (Injury, poisoning and procedural complications) | 3 | 1
Fracture (Injury, poisoning and procedural complications) | 5 | 5
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 1
Fractured coccyx (Injury, poisoning and procedural complications) | 1 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0
Haemarthrosis (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 7 | 7
Hip fracture (Injury, poisoning and procedural complications) | 1 | 3
Humerus fracture (Injury, poisoning and procedural complications) | 6 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 5 | 6
Lower limb fracture (Injury, poisoning and procedural complications) | 3 | 4
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 1
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 6 | 2
Rib fracture (Injury, poisoning and procedural complications) | 7 | 6
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 5 | 7
Traumatic fracture (Injury, poisoning and procedural complications) | 2 | 2
Ulna fracture (Injury, poisoning and procedural complications) | 2 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 18 | 7
Wrist fracture (Injury, poisoning and procedural complications) | 30 | 15
Food poisoning (Injury, poisoning and procedural complications) | 6 | 7
Animal bite (Injury, poisoning and procedural complications) | 0 | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 2
Excoriation (Injury, poisoning and procedural complications) | 10 | 9
Fall (Injury, poisoning and procedural complications) | 19 | 16
Injury (Injury, poisoning and procedural complications) | 0 | 2
Ligament injury (Injury, poisoning and procedural complications) | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Mouth injury (Injury, poisoning and procedural complications) | 2 | 2
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1
Perineal laceration (Injury, poisoning and procedural complications) | 0 | 1
Retinal detachment (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 3 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 10 | 13
Superficial injury of eye (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 4 | 1
Tooth injury (Injury, poisoning and procedural complications) | 1 | 1
Vascular injury (Injury, poisoning and procedural complications) | 1 | 1
Vena cava injury (Injury, poisoning and procedural complications) | 0 | 1
Vitreous detachment (Injury, poisoning and procedural complications) | 0 | 1
Deep vein thrombosis postoperative (Injury, poisoning and procedural complications) | 1 | 0
Device intolerance (Injury, poisoning and procedural complications) | 1 | 0
Implant tissue necrosis (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Postoperative thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 3 | 11
Seroma (Injury, poisoning and procedural complications) | 1 | 1
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 1
Biopsy lymph gland (Investigations) | 1 | 1
Angiogram (Investigations) | 1 | 0
Arteriogram coronary (Investigations) | 1 | 1
Blood pressure (Investigations) | 2 | 2
Blood pressure abnormal (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 1 | 0
Cardiac murmur (Investigations) | 1 | 0
Cardiovascular evaluation (Investigations) | 0 | 1
Catheterisation cardiac (Investigations) | 1 | 0
Echocardiogram (Investigations) | 0 | 1
Electrocardiogram (Investigations) | 3 | 2
Electrocardiogram abnormal (Investigations) | 0 | 2
Electrocardiogram ST segment depression (Investigations) | 0 | 1
Heart rate decreased (Investigations) | 0 | 1
Heart rate irregular (Investigations) | 1 | 1
Scan myocardial perfusion (Investigations) | 0 | 1
Ultrasound Doppler (Investigations) | 0 | 2
Venogram (Investigations) | 0 | 1
Gene mutation identification test positive (Investigations) | 1 | 0
Biopsy thyroid gland (Investigations) | 1 | 0
Thyroid function test abnormal (Investigations) | 0 | 1
Barium enema (Investigations) | 1 | 0
Barium swallow (Investigations) | 1 | 0
Biopsy colon abnormal (Investigations) | 1 | 0
Biopsy oesophagus (Investigations) | 0 | 1
Colonoscopy (Investigations) | 0 | 5
Endoscopy upper gastrointestinal tract (Investigations) | 2 | 5
Oesophagogastroscopy (Investigations) | 0 | 1
Sigmoidoscopy (Investigations) | 1 | 1
Ultrasound abdomen (Investigations) | 1 | 2
White blood cell count decreased (Investigations) | 1 | 0
Red blood cell count (Investigations) | 2 | 0
Biopsy liver (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 17 | 21
Ultrasound biliary tract (Investigations) | 0 | 1
Biopsy (Investigations) | 0 | 1
Computerised tomogram (Investigations) | 1 | 0
Endoscopy (Investigations) | 1 | 0
Imaging procedure (Investigations) | 1 | 0
Investigation (Investigations) | 2 | 0
Needle biopsy site unspecified normal (Investigations) | 1 | 0
Nuclear magnetic resonance imaging (Investigations) | 4 | 2
X-ray (Investigations) | 4 | 2
Free fatty acids increased (Investigations) | 0 | 1
Glucose tolerance test (Investigations) | 5 | 3
Arthroscopy (Investigations) | 6 | 7
Bone densitometry (Investigations) | 4 | 3
Bone density decreased (Investigations) | 56 | 42
Acoustic stimulation tests (Investigations) | 0 | 1
Brain scan normal (Investigations) | 0 | 1
Scan brain (Investigations) | 0 | 1
Body height decreased (Investigations) | 0 | 1
Body temperature increased (Investigations) | 4 | 1
Gastrointestinal examination (Investigations) | 1 | 1
Gynaecological examination (Investigations) | 1 | 1
Neurological examination (Investigations) | 1 | 0
Ophthalmological examination (Investigations) | 4 | 4
Orthopedic examination (Investigations) | 0 | 2
Weight decreased (Investigations) | 23 | 15
Weight increased (Investigations) | 126 | 133
Cystoscopy (Investigations) | 0 | 1
Ultrasound kidney (Investigations) | 2 | 1
Aspiration breast (Investigations) | 3 | 3
Biopsy breast (Investigations) | 8 | 12
Biopsy breast normal (Investigations) | 1 | 0
Biopsy cervix (Investigations) | 1 | 1
Biopsy endometrium (Investigations) | 2 | 7
Biopsy endometrium normal (Investigations) | 0 | 1
Biopsy testes normal (Investigations) | 0 | 1
Biopsy uterus (Investigations) | 0 | 3
Biopsy vagina (Investigations) | 0 | 1
Hysteroscopy (Investigations) | 4 | 16
Mammogram (Investigations) | 3 | 3
Mammogram abnormal (Investigations) | 0 | 1
Mammogram normal (Investigations) | 0 | 2
Smear cervix (Investigations) | 0 | 1
Smear cervix abnormal (Investigations) | 1 | 6
Ultrasound breast (Investigations) | 2 | 10
Ultrasound pelvis (Investigations) | 0 | 1
Ultrasound scan vagina (Investigations) | 0 | 4
Ultrasound uterus (Investigations) | 0 | 2
Chest X-ray (Investigations) | 1 | 1
Computerised tomogram thorax (Investigations) | 0 | 1
Laryngoscopy (Investigations) | 0 | 1
Sclerotherapy (Investigations) | 1 | 0
Serum ferritin increased (Investigations) | 1 | 0
Arrhythmia (Cardiac disorders) | 5 | 7
Atrial fibrillation (Cardiac disorders) | 5 | 5
Atrial flutter (Cardiac disorders) | 0 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 1
Bradyarrhythmia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 9 | 9
Cardiac discomfort (Cardiac disorders) | 1 | 0
Cardiac disorder (Cardiac disorders) | 2 | 1
Cardiovascular disorder (Cardiac disorders) | 2 | 1
Dizziness (Cardiac disorders) | 1 | 0
Dyspnoea (Cardiac disorders) | 0 | 2
Palpitations (Cardiac disorders) | 19 | 18
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Mitral valve prolapse (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 6 | 0
Angina unstable (Cardiac disorders) | 2 | 0
Chest pain (Cardiac disorders) | 14 | 15
Coronary artery disease (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 1
Endocarditis (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1
Cardiomegaly (Cardiac disorders) | 2 | 6
Cardiomyopathy (Cardiac disorders) | 2 | 0
Ventricular dysfunction (Cardiac disorders) | 0 | 1
Dressler's syndrome (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 1
Gastrointestinal angiodysplasia (Congenital, familial and genetic disorders) | 0 | 1
Heart disease congenital (Congenital, familial and genetic disorders) | 0 | 1
Cataract congenital (Congenital, familial and genetic disorders) | 0 | 1
Haemangioma of retina (Congenital, familial and genetic disorders) | 0 | 1
Osteopetrosis (Congenital, familial and genetic disorders) | 1 | 0
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 2 | 0
Basal cell naevus syndrome (Congenital, familial and genetic disorders) | 1 | 0
Keratosis follicular (Congenital, familial and genetic disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 3 | 3
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 2
Coagulopathy (Blood and lymphatic system disorders) | 1 | 2
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 4
Blood disorder (Blood and lymphatic system disorders) | 3 | 2
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Chronic lymphocytic leukaemia (Blood and lymphatic system disorders) | 1 | 0
Non-Hodgkin's lymphoma (Blood and lymphatic system disorders) | 0 | 1
Gammopathy (Blood and lymphatic system disorders) | 2 | 0
Multiple myeloma (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 2
Lymphoedema (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 4 | 4
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebral vasoconstriction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 2
Temporal arteritis (Nervous system disorders) | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 3 | 1
Anosmia (Nervous system disorders) | 2 | 0
Cranial nerve paralysis (Nervous system disorders) | 0 | 1
Facial palsy (Nervous system disorders) | 1 | 3
Facial spasm (Nervous system disorders) | 0 | 1
Neuritis cranial (Nervous system disorders) | 0 | 1
Optic neuritis (Nervous system disorders) | 0 | 1
VIth nerve paralysis (Nervous system disorders) | 0 | 1
Multiple sclerosis (Nervous system disorders) | 1 | 4
Headache (Nervous system disorders) | 82 | 61
Migraine (Nervous system disorders) | 10 | 10
Migraine with aura (Nervous system disorders) | 1 | 0
Tension headache (Nervous system disorders) | 1 | 0
Amnesia (Nervous system disorders) | 27 | 28
Cognitive disorder (Nervous system disorders) | 3 | 0
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0
Dementia of the Alzheimer's type, with depressed mood (Nervous system disorders) | 1 | 0
Disturbance in attention (Nervous system disorders) | 2 | 4
Memory impairment (Nervous system disorders) | 1 | 1
Essential tremor (Nervous system disorders) | 0 | 1
Parkinsonism (Nervous system disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 2 | 1
Spastic paralysis (Nervous system disorders) | 0 | 1
Torticollis (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 2 | 10
Ageusia (Nervous system disorders) | 0 | 1
Analgesia (Nervous system disorders) | 0 | 1
Aphonia (Nervous system disorders) | 2 | 6
Balance disorder (Nervous system disorders) | 35 | 35
Confusional state (Nervous system disorders) | 4 | 2
Coordination abnormal (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 7 | 8
Dizziness postural (Nervous system disorders) | 1 | 0
Dysaesthesia (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 11 | 3
Hypoaesthesia (Nervous system disorders) | 10 | 10
Lethargy (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 5 | 4
Neurological symptom (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 43 | 23
Presyncope (Nervous system disorders) | 1 | 1
Restless legs syndrome (Nervous system disorders) | 2 | 3
Sensory disturbance (Nervous system disorders) | 8 | 1
Somnolence (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Vertigo (Nervous system disorders) | 15 | 17
Muscle rigidity (Nervous system disorders) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 35 | 13
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1
Nerve compression (Nervous system disorders) | 4 | 2
Neuropathy peripheral (Nervous system disorders) | 17 | 14
Convulsion (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 3 | 0
Insomnia (Nervous system disorders) | 3 | 0
Narcolepsy (Nervous system disorders) | 0 | 3
Radiculopathy (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 10 | 11
Cataract (Eye disorders) | 77 | 64
Cataract congenital (Eye disorders) | 0 | 1
Cataract diabetic (Eye disorders) | 1 | 0
Cataract nuclear (Eye disorders) | 1 | 0
Entropion (Eye disorders) | 0 | 1
Corneal disorder (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 35 | 49
Eye disorder (Eye disorders) | 38 | 35
Eye pain (Eye disorders) | 8 | 5
Eyelid disorder (Eye disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 12 | 7
Vitreous disorder (Eye disorders) | 0 | 1
Borderline glaucoma (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 21 | 15
Ocular hypertension (Eye disorders) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 1
Eye haemorrhage (Eye disorders) | 1 | 2
Blepharitis (Eye disorders) | 7 | 3
Conjunctivitis (Eye disorders) | 5 | 6
Episcleritis (Eye disorders) | 0 | 1
Eye irritation (Eye disorders) | 9 | 8
Ocular hyperaemia (Eye disorders) | 2 | 3
Haemangioma of retina (Eye disorders) | 0 | 1
Blepharospasm (Eye disorders) | 0 | 3
Macular degeneration (Eye disorders) | 8 | 5
Macular hole (Eye disorders) | 2 | 1
Retinal detachment (Eye disorders) | 4 | 4
Retinal tear (Eye disorders) | 0 | 1
Vitreous detachment (Eye disorders) | 6 | 4
Diabetic retinopathy (Eye disorders) | 3 | 0
Retinal artery occlusion (Eye disorders) | 3 | 0
Retinal vein occlusion (Eye disorders) | 1 | 1
Retinal vein thrombosis (Eye disorders) | 1 | 0
Blindness (Eye disorders) | 0 | 1
Diplopia (Eye disorders) | 1 | 2
Myopia (Eye disorders) | 3 | 1
Vision blurred (Eye disorders) | 12 | 18
Visual acuity reduced (Eye disorders) | 40 | 42
Visual impairment (Eye disorders) | 11 | 14
Cholesteatoma (Ear and labyrinth disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 2 | 3
Deafness (Ear and labyrinth disorders) | 6 | 5
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 7 | 4
Vertigo (Ear and labyrinth disorders) | 3 | 1
Mastoid disorder (Ear and labyrinth disorders) | 1 | 0
Mastoiditis (Ear and labyrinth disorders) | 1 | 0
Middle ear adhesions (Ear and labyrinth disorders) | 0 | 1
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 4
Femoral hernia (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 6 | 5
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Lumbar hernia (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 2 | 3
Anal pruritus (Gastrointestinal disorders) | 1 | 0
Anorectal disorder (Gastrointestinal disorders) | 0 | 1
Anorectal squamous cell metaplasia (Gastrointestinal disorders) | 1 | 0
Rectal prolapse (Gastrointestinal disorders) | 3 | 1
Anal polyp (Gastrointestinal disorders) | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 1
Gastric polyps (Gastrointestinal disorders) | 2 | 0
Intestinal polyp (Gastrointestinal disorders) | 0 | 1
Rectal polyp (Gastrointestinal disorders) | 0 | 1
Gingival disorder (Gastrointestinal disorders) | 8 | 5
Gingivitis (Gastrointestinal disorders) | 1 | 0
Poor dental condition (Gastrointestinal disorders) | 1 | 0
Tooth fracture (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 2
Diverticulitis (Gastrointestinal disorders) | 7 | 9
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 2 | 1
Barrett's oesophagus (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 1
Gastric mucosal hypertrophy (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 4 | 12
Oesophageal disorder (Gastrointestinal disorders) | 1 | 2
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 9
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 3
Colitis ischaemic (Gastrointestinal disorders) | 1 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 12 | 13
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1
Inflammatory bowel disease (Gastrointestinal disorders) | 0 | 2
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Proctocolitis (Gastrointestinal disorders) | 0 | 2
Reflux oesophagitis (Gastrointestinal disorders) | 17 | 18
Change of bowel habit (Gastrointestinal disorders) | 5 | 2
Constipation (Gastrointestinal disorders) | 24 | 42
Diarrhoea (Gastrointestinal disorders) | 20 | 18
Duodenogastric reflux (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2
Irritable bowel syndrome (Gastrointestinal disorders) | 5 | 3
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 15 | 11
Abdominal mass (Gastrointestinal disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 33 | 48
Dyspepsia (Gastrointestinal disorders) | 25 | 24
Dysphagia (Gastrointestinal disorders) | 3 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 9 | 10
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 57 | 51
Pelvic pain (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 9 | 7
Gallstone ileus (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 6 | 7
Coeliac disease (Gastrointestinal disorders) | 2 | 0
Anal cancer (Gastrointestinal disorders) | 1 | 0
Rectal cancer (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 3 | 7
Oral pain (Gastrointestinal disorders) | 2 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 0
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 25 | 16
Dry throat (Gastrointestinal disorders) | 1 | 0
Lip dry (Gastrointestinal disorders) | 1 | 0
Salivary gland cyst (Gastrointestinal disorders) | 0 | 1
Salivary gland disorder (Gastrointestinal disorders) | 0 | 1
Ageusia (Gastrointestinal disorders) | 0 | 1
Glossitis (Gastrointestinal disorders) | 0 | 2
Tongue disorder (Gastrointestinal disorders) | 0 | 1
Bladder disorder (Renal and urinary disorders) | 1 | 0
Bladder prolapse (Renal and urinary disorders) | 0 | 1
Calculus bladder (Renal and urinary disorders) | 0 | 2
Chromaturia (Renal and urinary disorders) | 1 | 0
Cystitis (Renal and urinary disorders) | 1 | 1
Dysuria (Renal and urinary disorders) | 2 | 6
Haematuria (Renal and urinary disorders) | 2 | 1
Haemorrhage urinary tract (Renal and urinary disorders) | 1 | 0
Micturition disorder (Renal and urinary disorders) | 7 | 16
Micturition urgency (Renal and urinary disorders) | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 3 | 0
Nocturia (Renal and urinary disorders) | 1 | 1
Pollakiuria (Renal and urinary disorders) | 6 | 10
Polyuria (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 2
Renal cyst (Renal and urinary disorders) | 1 | 0
Renal disorder (Renal and urinary disorders) | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Renal tubular acidosis (Renal and urinary disorders) | 1 | 0
Stress urinary incontinence (Renal and urinary disorders) | 1 | 3
Urethral stenosis (Renal and urinary disorders) | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 6 | 15
Urinary tract infection (Renal and urinary disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 4
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 80 | 93
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 | 1
Basal cell carcinoma (Skin and subcutaneous tissue disorders) | 0 | 2
Basal cell naevus syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 2 | 2
Bowen's disease (Skin and subcutaneous tissue disorders) | 1 | 0
Cellulitis (Skin and subcutaneous tissue disorders) | 2 | 4
Dermal cyst (Skin and subcutaneous tissue disorders) | 6 | 5
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 27 | 28
Eczema (Skin and subcutaneous tissue disorders) | 6 | 18
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 5 | 3
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 1 | 0
Hair disorder (Skin and subcutaneous tissue disorders) | 5 | 11
Hirsutism (Skin and subcutaneous tissue disorders) | 6 | 12
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 25 | 18
Lichen planus (Skin and subcutaneous tissue disorders) | 1 | 0
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 1 | 3
Morphoea (Skin and subcutaneous tissue disorders) | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 6 | 13
Night sweats (Skin and subcutaneous tissue disorders) | 310 | 341
Onychoclasis (Skin and subcutaneous tissue disorders) | 6 | 16
Periorbital oedema (Skin and subcutaneous tissue disorders) | 2 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 2 | 2
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 2 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 22 | 38
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 6 | 3
Rash (Skin and subcutaneous tissue disorders) | 26 | 37
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Rash scarlatiniform (Skin and subcutaneous tissue disorders) | 1 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 6
Scar (Skin and subcutaneous tissue disorders) | 1 | 0
Scar pain (Skin and subcutaneous tissue disorders) | 1 | 4
Skin atrophy (Skin and subcutaneous tissue disorders) | 1 | 0
Skin cancer (Skin and subcutaneous tissue disorders) | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 12 | 12
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 3 | 2
Skin swelling (Skin and subcutaneous tissue disorders) | 2 | 6
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 | 1
Skin warm (Skin and subcutaneous tissue disorders) | 1 | 0
Superficial spreading melanoma stage unspecified (Skin and subcutaneous tissue disorders) | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 2
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 6 | 11
Varicella (Skin and subcutaneous tissue disorders) | 1 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 2 | 0
Bone erosion (Musculoskeletal and connective tissue disorders) | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Jaw disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteitis deformans (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 11 | 4
Osteoporosis (Musculoskeletal and connective tissue disorders) | 106 | 71
Osteoporosis postmenopausal (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 | 1
CREST syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Morphoea (Musculoskeletal and connective tissue disorders) | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 5 | 2
Scleroderma (Musculoskeletal and connective tissue disorders) | 1 | 0
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 2 | 1
Ankle fracture (Musculoskeletal and connective tissue disorders) | 0 | 2
Clavicle fracture (Musculoskeletal and connective tissue disorders) | 0 | 2
Fibula fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Foot fracture (Musculoskeletal and connective tissue disorders) | 2 | 2
Forearm fracture (Musculoskeletal and connective tissue disorders) | 3 | 0
Fractured coccyx (Musculoskeletal and connective tissue disorders) | 1 | 0
Hand fracture (Musculoskeletal and connective tissue disorders) | 0 | 2
Hip fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Humerus fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Lower limb fracture (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 3 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 1
Radius fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Rib fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal fracture (Musculoskeletal and connective tissue disorders) | 2 | 2
Thoracic vertebral fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Upper limb fracture (Musculoskeletal and connective tissue disorders) | 2 | 0
Wrist fracture (Musculoskeletal and connective tissue disorders) | 3 | 1
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 842 | 748
Arthritis (Musculoskeletal and connective tissue disorders) | 52 | 50
Arthritis bacterial (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis infective (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 11 | 9
Floating patella (Musculoskeletal and connective tissue disorders) | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint dislocation (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 2 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 74 | 37
Joint swelling (Musculoskeletal and connective tissue disorders) | 18 | 17
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 3 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 67 | 53
Palindromic rheumatism (Musculoskeletal and connective tissue disorders) | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 9 | 4
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 15 | 12
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Senile ankylosing vertebral hyperostosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 6
Spondylitis (Musculoskeletal and connective tissue disorders) | 2 | 3
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 26 | 108
Myalgia (Musculoskeletal and connective tissue disorders) | 124 | 106
Periodic limb movement disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Torticollis (Musculoskeletal and connective tissue disorders) | 1 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 3 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 6 | 7
Lumbar spine flattening (Musculoskeletal and connective tissue disorders) | 0 | 1
Sciatica (Musculoskeletal and connective tissue disorders) | 0 | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Back disorder (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 82 | 101
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 2 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 100 | 95
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 19 | 18
Neck mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 101 | 80
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 4 | 5
Bunion (Musculoskeletal and connective tissue disorders) | 1 | 3
Bursitis (Musculoskeletal and connective tissue disorders) | 2 | 11
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 2
Cartilage injury (Musculoskeletal and connective tissue disorders) | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 18 | 8
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 10 | 4
Breast cancer (Musculoskeletal and connective tissue disorders) | 3 | 6
Adrenal adenoma (Endocrine disorders) | 1 | 0
Adrenal carcinoma (Endocrine disorders) | 0 | 1
Adrenal disorder (Endocrine disorders) | 0 | 1
Adrenal mass (Endocrine disorders) | 0 | 1
Diabetes mellitus (Endocrine disorders) | 2 | 0
Type 2 diabetes mellitus (Endocrine disorders) | 0 | 4
Hypoparathyroidism (Endocrine disorders) | 0 | 1
Parathyroid disorder (Endocrine disorders) | 0 | 1
Goitre (Endocrine disorders) | 6 | 5
Hyperthyroidism (Endocrine disorders) | 3 | 0
Hypothyroidism (Endocrine disorders) | 12 | 16
Thyroid cyst (Endocrine disorders) | 2 | 2
Thyroid disorder (Endocrine disorders) | 2 | 2
Renal tubular acidosis (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 10 | 6
Increased appetite (Metabolism and nutrition disorders) | 2 | 0
Weight fluctuation (Metabolism and nutrition disorders) | 6 | 2
Bone metabolism disorder (Metabolism and nutrition disorders) | 0 | 1
Osteopenia (Metabolism and nutrition disorders) | 1 | 0
Osteoporosis (Metabolism and nutrition disorders) | 4 | 2
Diabetic foot (Metabolism and nutrition disorders) | 1 | 1
Fluid retention (Metabolism and nutrition disorders) | 3 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 21 | 13
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 4
Haemochromatosis (Metabolism and nutrition disorders) | 0 | 2
Iron deficiency anaemia (Metabolism and nutrition disorders) | 2 | 3
Iron overload (Metabolism and nutrition disorders) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 47 | 11
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 | 8
Goitre (Metabolism and nutrition disorders) | 1 | 0
Hypothyroidism (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 2
Folate deficiency (Metabolism and nutrition disorders) | 0 | 1
Multi-vitamin deficiency (Metabolism and nutrition disorders) | 1 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1
Vitamin B6 deficiency (Metabolism and nutrition disorders) | 1 | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 2
Subacute sclerosing panencephalitis (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 5 | 2
Breast cellulitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 2
Folliculitis (Infections and infestations) | 0 | 1
Helicobacter gastritis (Infections and infestations) | 1 | 0
Helicobacter infection (Infections and infestations) | 2 | 0
Lyme disease (Infections and infestations) | 0 | 3
Staphylococcal infection (Infections and infestations) | 0 | 1
Fungal infection (Infections and infestations) | 3 | 3
Oral candidiasis (Infections and infestations) | 0 | 3
Pneumonia cryptococcal (Infections and infestations) | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 9 | 42
Acute sinusitis (Infections and infestations) | 1 | 3
Arthritis infective (Infections and infestations) | 1 | 1
Breast abscess (Infections and infestations) | 0 | 1
Bronchiectasis (Infections and infestations) | 0 | 2
Chronic sinusitis (Infections and infestations) | 3 | 3
Cystitis (Infections and infestations) | 14 | 14
Diverticulitis (Infections and infestations) | 4 | 5
Eye infection (Infections and infestations) | 1 | 2
Furuncle (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 2
Hordeolum (Infections and infestations) | 0 | 1
Incision site infection (Infections and infestations) | 0 | 1
Labyrinthitis (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 1 | 2
Lower respiratory tract infection (Infections and infestations) | 5 | 14
Lung infection (Infections and infestations) | 1 | 0
Mastitis (Infections and infestations) | 2 | 0
Otitis externa (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 4 | 4
Paronychia (Infections and infestations) | 0 | 3
Pharyngitis (Infections and infestations) | 2 | 7
Pneumonia (Infections and infestations) | 5 | 0
Post procedural infection (Infections and infestations) | 3 | 3
Respiratory tract infection (Infections and infestations) | 1 | 1
Rhinitis (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 1 | 2
Sialoadenitis (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 2 | 0
Skin infection (Infections and infestations) | 1 | 4
Tonsillitis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 5 | 7
Upper respiratory tract infection (Infections and infestations) | 6 | 5
Urinary tract infection (Infections and infestations) | 23 | 32
Wound infection (Infections and infestations) | 1 | 1
Mycobacterial infection (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Toxoplasmosis (Infections and infestations) | 1 | 0
Hepatitis viral (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 11 | 13
Influenza (Infections and infestations) | 2 | 14
Post viral fatigue syndrome (Infections and infestations) | 0 | 2
Vestibular neuronitis (Infections and infestations) | 1 | 2
Viral infection (Infections and infestations) | 7 | 8
Accelerated hypertension (Vascular disorders) | 1 | 0
Aneurysm (Vascular disorders) | 0 | 1
Angina unstable (Vascular disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 1
Carotid artery occlusion (Vascular disorders) | 0 | 1
Carotid artery stenosis (Vascular disorders) | 1 | 0
Cerebrovascular accident (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 2
Coronary artery disease (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 5 | 3
Dizziness (Vascular disorders) | 0 | 1
Embolism (Vascular disorders) | 2 | 5
Epistaxis (Vascular disorders) | 0 | 1
Essential hypertension (Vascular disorders) | 68 | 54
Femoral artery aneurysm (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 4 | 8
Haemorrhage intracranial (Vascular disorders) | 0 | 1
Hot flush (Vascular disorders) | 161 | 184
Hypertension (Vascular disorders) | 28 | 22
Hypotension (Vascular disorders) | 2 | 3
Ischaemia (Vascular disorders) | 1 | 0
Ischaemic stroke (Vascular disorders) | 1 | 2
Lymphoedema (Vascular disorders) | 4 | 8
Malignant hypertension (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Peripheral coldness (Vascular disorders) | 3 | 3
Peripheral vascular disorder (Vascular disorders) | 2 | 1
Phlebitis (Vascular disorders) | 3 | 7
Postmenopausal haemorrhage (Vascular disorders) | 0 | 1
Presyncope (Vascular disorders) | 1 | 0
Pulmonary embolism (Vascular disorders) | 3 | 2
Spider vein (Vascular disorders) | 1 | 0
Syncope (Vascular disorders) | 1 | 2
Temporal arteritis (Vascular disorders) | 0 | 2
Thrombophlebitis superficial (Vascular disorders) | 1 | 6
Thrombosis (Vascular disorders) | 1 | 0
Transient ischaemic attack (Vascular disorders) | 7 | 2
Varicose ulceration (Vascular disorders) | 0 | 1
Varicose vein (Vascular disorders) | 7 | 9
Vasculitis (Vascular disorders) | 0 | 1
Venous insufficiency (Vascular disorders) | 3 | 0
Venous thrombosis (Vascular disorders) | 0 | 1
Abscess drainage (Surgical and medical procedures) | 1 | 0
Acupuncture (Surgical and medical procedures) | 0 | 1
Adrenal gland operation (Surgical and medical procedures) | 0 | 1
Anal polypectomy (Surgical and medical procedures) | 0 | 1
Angioplasty (Surgical and medical procedures) | 2 | 2
Ankle operation (Surgical and medical procedures) | 1 | 0
Aortic valve replacement (Surgical and medical procedures) | 1 | 0
Appendicectomy (Surgical and medical procedures) | 0 | 1
Arterial stent insertion (Surgical and medical procedures) | 1 | 0
Arthroscopic surgery (Surgical and medical procedures) | 0 | 1
Bladder operation (Surgical and medical procedures) | 0 | 1
Bone lesion excision (Surgical and medical procedures) | 1 | 0
Bone operation (Surgical and medical procedures) | 0 | 1
Breast cyst drainage (Surgical and medical procedures) | 1 | 2
Breast lump removal (Surgical and medical procedures) | 1 | 3
Breast reconstruction (Surgical and medical procedures) | 1 | 0
Bunion operation (Surgical and medical procedures) | 6 | 8
Cancer surgery (Surgical and medical procedures) | 0 | 1
Cardiac ablation (Surgical and medical procedures) | 0 | 2
Cardiac operation (Surgical and medical procedures) | 1 | 0
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 | 0
Cardiac resynchronisation therapy (Surgical and medical procedures) | 1 | 0
Cardioversion (Surgical and medical procedures) | 1 | 0
Carpal tunnel decompression (Surgical and medical procedures) | 13 | 3
Cataract operation (Surgical and medical procedures) | 18 | 26
Cervical polypectomy (Surgical and medical procedures) | 1 | 1
Chemotherapy (Surgical and medical procedures) | 1 | 2
Chiropractic (Surgical and medical procedures) | 1 | 0
Cholecystectomy (Surgical and medical procedures) | 9 | 7
Colon operation (Surgical and medical procedures) | 1 | 0
Colon polypectomy (Surgical and medical procedures) | 3 | 6
Colonoscopy (Surgical and medical procedures) | 1 | 4
Colostomy (Surgical and medical procedures) | 0 | 2
Colporrhaphy (Surgical and medical procedures) | 0 | 1
Coronary artery bypass (Surgical and medical procedures) | 1 | 1
Cyst removal (Surgical and medical procedures) | 1 | 0
Debridement (Surgical and medical procedures) | 1 | 0
Dental care (Surgical and medical procedures) | 1 | 0
Dental implantation (Surgical and medical procedures) | 0 | 1
Dupuytren's contracture operation (Surgical and medical procedures) | 0 | 1
Ear operation (Surgical and medical procedures) | 0 | 1
Elbow operation (Surgical and medical procedures) | 1 | 0
Elective surgery (Surgical and medical procedures) | 1 | 0
Emergency care (Surgical and medical procedures) | 1 | 3
Endocervical curettage (Surgical and medical procedures) | 0 | 1
Ethmoid sinus surgery (Surgical and medical procedures) | 0 | 1
Eye operation (Surgical and medical procedures) | 3 | 3
Foot operation (Surgical and medical procedures) | 2 | 2
Gallbladder operation (Surgical and medical procedures) | 0 | 1
Haemorrhoid operation (Surgical and medical procedures) | 0 | 1
Hand repair operation (Surgical and medical procedures) | 0 | 1
Heart valve replacement (Surgical and medical procedures) | 0 | 2
Hernia repair (Surgical and medical procedures) | 1 | 0
High frequency ablation (Surgical and medical procedures) | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 14 | 10
Hip surgery (Surgical and medical procedures) | 6 | 4
Hospitalisation (Surgical and medical procedures) | 3 | 3
Hysterectomy (Surgical and medical procedures) | 4 | 17
Ileostomy (Surgical and medical procedures) | 0 | 1
Incisional hernia repair (Surgical and medical procedures) | 0 | 2
Inguinal hernia repair (Surgical and medical procedures) | 0 | 1
Intervertebral disc operation (Surgical and medical procedures) | 1 | 0
Intestinal resection (Surgical and medical procedures) | 0 | 1
Intraocular lens implant (Surgical and medical procedures) | 1 | 0
Intra-uterine contraceptive device (Surgical and medical procedures) | 0 | 1
Jaw operation (Surgical and medical procedures) | 1 | 0
Joint manipulation (Surgical and medical procedures) | 0 | 1
Joint surgery (Surgical and medical procedures) | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 12 | 13
Knee operation (Surgical and medical procedures) | 8 | 3
Large intestine operation (Surgical and medical procedures) | 0 | 1
Laryngeal polypectomy (Surgical and medical procedures) | 0 | 1
Lesion excision (Surgical and medical procedures) | 1 | 0
Limb operation (Surgical and medical procedures) | 1 | 3
Lipoma excision (Surgical and medical procedures) | 0 | 7
Local anaesthesia (Surgical and medical procedures) | 3 | 0
Lung lobectomy (Surgical and medical procedures) | 2 | 1
Lymphadenectomy (Surgical and medical procedures) | 0 | 1
Mammoplasty (Surgical and medical procedures) | 3 | 4
Mastectomy (Surgical and medical procedures) | 2 | 4
Meningioma surgery (Surgical and medical procedures) | 1 | 0
Meniscus removal (Surgical and medical procedures) | 2 | 3
Mitral valve replacement (Surgical and medical procedures) | 0 | 1
Mole excision (Surgical and medical procedures) | 0 | 1
Muscle operation (Surgical and medical procedures) | 1 | 0
Nail operation (Surgical and medical procedures) | 2 | 0
Nasal operation (Surgical and medical procedures) | 0 | 1
Nephrectomy (Surgical and medical procedures) | 1 | 0
Nerve block (Surgical and medical procedures) | 0 | 1
Oophorectomy (Surgical and medical procedures) | 0 | 3
Oophorectomy bilateral (Surgical and medical procedures) | 2 | 5
Open reduction of fracture (Surgical and medical procedures) | 0 | 1
Ovarian cystectomy (Surgical and medical procedures) | 3 | 1
Parathyroidectomy (Surgical and medical procedures) | 2 | 1
Pelvic floor repair (Surgical and medical procedures) | 1 | 4
Physiotherapy (Surgical and medical procedures) | 0 | 1
Plastic surgery (Surgical and medical procedures) | 1 | 1
Polypectomy (Surgical and medical procedures) | 1 | 12
Prolapse repair (Surgical and medical procedures) | 1 | 0
Prosthesis implantation (Surgical and medical procedures) | 1 | 0
Radical mastectomy (Surgical and medical procedures) | 1 | 0
Radiotherapy (Surgical and medical procedures) | 1 | 2
Renal cyst excision (Surgical and medical procedures) | 1 | 0
Retinal laser coagulation (Surgical and medical procedures) | 2 | 1
Retinal operation (Surgical and medical procedures) | 0 | 2
Salpingectomy (Surgical and medical procedures) | 0 | 2
Salpingo-oophorectomy (Surgical and medical procedures) | 0 | 1
Salpingo-oophorectomy bilateral (Surgical and medical procedures) | 1 | 2
Sclerotherapy (Surgical and medical procedures) | 1 | 0
Shoulder arthroplasty (Surgical and medical procedures) | 0 | 1
Shoulder operation (Surgical and medical procedures) | 6 | 3
Simple mastectomy (Surgical and medical procedures) | 1 | 0
Sinus operation (Surgical and medical procedures) | 0 | 1
Skin graft (Surgical and medical procedures) | 1 | 0
Skin lesion excision (Surgical and medical procedures) | 5 | 3
Skin neoplasm excision (Surgical and medical procedures) | 2 | 4
Spinal decompression (Surgical and medical procedures) | 1 | 2
Spinal laminectomy (Surgical and medical procedures) | 1 | 0
Spinal operation (Surgical and medical procedures) | 2 | 2
Stent placement (Surgical and medical procedures) | 2 | 0
Steroid therapy (Surgical and medical procedures) | 1 | 0
Surgery (Surgical and medical procedures) | 4 | 4
Tendon operation (Surgical and medical procedures) | 1 | 0
Tendon sheath lesion excision (Surgical and medical procedures) | 1 | 0
Therapeutic skin care topical (Surgical and medical procedures) | 0 | 1
Thoracotomy (Surgical and medical procedures) | 0 | 1
Thyroid operation (Surgical and medical procedures) | 3 | 1
Thyroidectomy (Surgical and medical procedures) | 1 | 3
Toe amputation (Surgical and medical procedures) | 0 | 1
Toe operation (Surgical and medical procedures) | 1 | 0
Tooth extraction (Surgical and medical procedures) | 2 | 6
Trabeculectomy (Surgical and medical procedures) | 1 | 0
Transfusion (Surgical and medical procedures) | 1 | 0
Tumour excision (Surgical and medical procedures) | 0 | 1
Umbilical hernia repair (Surgical and medical procedures) | 0 | 1
Uterine cervix dilation procedure (Surgical and medical procedures) | 1 | 0
Uterine cystectomy (Surgical and medical procedures) | 0 | 1
Uterine dilation and curettage (Surgical and medical procedures) | 3 | 4
Uterine polypectomy (Surgical and medical procedures) | 3 | 0
Uterine prolapse repair (Surgical and medical procedures) | 1 | 0
Varicose vein operation (Surgical and medical procedures) | 1 | 0
Venous ligation (Surgical and medical procedures) | 1 | 2
Venous operation (Surgical and medical procedures) | 0 | 1
Vocal cordectomy (Surgical and medical procedures) | 0 | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 11
Breast cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 8
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anal polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric polyps (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Colorectal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Focal nodular hyperplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Adenoid cystic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Recurrent cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intracranial meningioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Genital cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervical polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Degeneration of uterine fibroid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Uterine cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 6
Uterine polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Vaginal polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Vulval polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Vulval neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nasal polyps (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenosquamous cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lung carcinoma cell type unspecified stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 9
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Asthma (Immune system disorders) | 2 | 0
Drug hypersensitivity (Immune system disorders) | 5 | 0
Hypersensitivity (Immune system disorders) | 3 | 10
Multiple allergies (Immune system disorders) | 1 | 0
Antiphospholipid syndrome (Immune system disorders) | 0 | 1
Polymyalgia rheumatica (Immune system disorders) | 1 | 1
Rheumatoid arthritis (Immune system disorders) | 0 | 1
Polyarteritis nodosa (Immune system disorders) | 0 | 1
Temporal arteritis (Immune system disorders) | 0 | 1
Bereavement (Social circumstances) | 0 | 1
Ex-tobacco user (Social circumstances) | 0 | 1
Pyrexia (General disorders) | 3 | 6
Asthenia (General disorders) | 23 | 25
Axillary pain (General disorders) | 0 | 1
Chest discomfort (General disorders) | 0 | 2
Chest pain (General disorders) | 4 | 6
Chills (General disorders) | 0 | 1
Disease recurrence (General disorders) | 0 | 1
Facial pain (General disorders) | 2 | 0
Fatigue (General disorders) | 1 | 2
Gait disturbance (General disorders) | 1 | 0
Hernia (General disorders) | 2 | 2
Hot flush (General disorders) | 19 | 14
Inflammation (General disorders) | 1 | 0
Influenza like illness (General disorders) | 0 | 1
Irritability (General disorders) | 6 | 1
Lethargy (General disorders) | 0 | 1
Malaise (General disorders) | 165 | 177
Night sweats (General disorders) | 5 | 3
Oedema (General disorders) | 21 | 28
Oedema peripheral (General disorders) | 18 | 9
Pain (General disorders) | 1 | 2
Polyp (General disorders) | 2 | 6
Thirst (General disorders) | 1 | 1
Adverse drug reaction (General disorders) | 0 | 1
Adverse reaction (General disorders) | 2 | 0
Cyst (General disorders) | 2 | 2
Dysplasia (General disorders) | 0 | 1
Fat necrosis (General disorders) | 2 | 1
Fibrosis (General disorders) | 6 | 3
Hyperplasia (General disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 2
Amnesia (Psychiatric disorders) | 2 | 0
Aggression (Psychiatric disorders) | 0 | 1
Alcohol problem (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 15 | 22
Bipolar I disorder (Psychiatric disorders) | 0 | 1
Cognitive disorder (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 67 | 70
Eating disorder (Psychiatric disorders) | 0 | 1
Emotional disorder (Psychiatric disorders) | 27 | 36
Hallucination (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 109 | 93
Loss of libido (Psychiatric disorders) | 10 | 12
Mental disorder (Psychiatric disorders) | 2 | 3
Nervousness (Psychiatric disorders) | 3 | 2
Neurosis (Psychiatric disorders) | 0 | 5
Nightmare (Psychiatric disorders) | 1 | 2
Personality disorder (Psychiatric disorders) | 3 | 0
Phobia (Psychiatric disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 2 | 3
Sleep disorder (Psychiatric disorders) | 1 | 0
Somnolence (Psychiatric disorders) | 1 | 0
Stress (Psychiatric disorders) | 4 | 5
Suicidal ideation (Psychiatric disorders) | 1 | 0
Adnexa uteri pain (Reproductive system and breast disorders) | 1 | 3
Arthritis climacteric (Reproductive system and breast disorders) | 0 | 1
Benign breast neoplasm (Reproductive system and breast disorders) | 0 | 1
Breast abscess (Reproductive system and breast disorders) | 0 | 1
Breast calcifications (Reproductive system and breast disorders) | 4 | 4
Breast cancer in situ (Reproductive system and breast disorders) | 1 | 3
Breast cancer metastatic (Reproductive system and breast disorders) | 1 | 0
Breast cancer recurrent (Reproductive system and breast disorders) | 1 | 0
Breast cyst (Reproductive system and breast disorders) | 10 | 7
Breast discharge (Reproductive system and breast disorders) | 6 | 5
Breast discomfort (Reproductive system and breast disorders) | 3 | 0
Breast disorder (Reproductive system and breast disorders) | 7 | 18
Breast hyperplasia (Reproductive system and breast disorders) | 2 | 1
Breast infection (Reproductive system and breast disorders) | 1 | 0
Breast necrosis (Reproductive system and breast disorders) | 0 | 1
Breast pain (Reproductive system and breast disorders) | 70 | 66
Breast swelling (Reproductive system and breast disorders) | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 2 | 0
Cervical polyp (Reproductive system and breast disorders) | 2 | 11
Cystocele (Reproductive system and breast disorders) | 1 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Dyspareunia (Reproductive system and breast disorders) | 11 | 11
Endometrial disorder (Reproductive system and breast disorders) | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 18
Endometrial hypertrophy (Reproductive system and breast disorders) | 2 | 34
Endometriosis (Reproductive system and breast disorders) | 1 | 1
Fibrocystic breast disease (Reproductive system and breast disorders) | 4 | 8
Galactorrhoea (Reproductive system and breast disorders) | 1 | 2
Gynaecomastia (Reproductive system and breast disorders) | 2 | 0
Hot flush (Reproductive system and breast disorders) | 815 | 898
Intraductal papilloma of breast (Reproductive system and breast disorders) | 1 | 0
Mastitis (Reproductive system and breast disorders) | 3 | 0
Menopausal symptoms (Reproductive system and breast disorders) | 1 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 13 | 20
Night sweats (Reproductive system and breast disorders) | 70 | 74
Nipple disorder (Reproductive system and breast disorders) | 0 | 1
Nipple pain (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 10 | 9
Ovarian mass (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Perineal pain (Reproductive system and breast disorders) | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 13 | 12
Premenstrual syndrome (Reproductive system and breast disorders) | 0 | 1
Sexual dysfunction (Reproductive system and breast disorders) | 1 | 2
Uterine atrophy (Reproductive system and breast disorders) | 1 | 0
Uterine cyst (Reproductive system and breast disorders) | 0 | 1
Uterine fibrosis (Reproductive system and breast disorders) | 1 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1
Uterine leiomyoma (Reproductive system and breast disorders) | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 9 | 25
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1
Uterine spasm (Reproductive system and breast disorders) | 1 | 3
Vaginal cyst (Reproductive system and breast disorders) | 1 | 2
Vaginal discharge (Reproductive system and breast disorders) | 31 | 140
Vaginal disorder (Reproductive system and breast disorders) | 20 | 22
Vaginal haemorrhage (Reproductive system and breast disorders) | 32 | 78
Vaginal inflammation (Reproductive system and breast disorders) | 0 | 2
Vaginal polyp (Reproductive system and breast disorders) | 1 | 2
Vaginal prolapse (Reproductive system and breast disorders) | 8 | 11
Vaginal swelling (Reproductive system and breast disorders) | 0 | 1
Vulval abscess (Reproductive system and breast disorders) | 0 | 1
Vulval neoplasm (Reproductive system and breast disorders) | 1 | 0
Vulval polyp (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 201 | 166
Vulvovaginal pain (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 19 | 47
Asthma (Respiratory, thoracic and mediastinal disorders) | 10 | 12
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Chest discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chest pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 24
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 | 30
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lobar pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Lower respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 22 | 53
Lung cancer metastatic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Multifocal micronodular pneumocyte hyperplasia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pertussis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 24 | 25
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tonsillitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 4 | 8
Gallbladder disorder (Hepatobiliary disorders) | 1 | 0
Haemochromatosis (Hepatobiliary disorders) | 0 | 2
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 3
Liver disorder (Hepatobiliary disorders) | 3 | 3
Hepatobiliary carcinoma in situ (Hepatobiliary disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
This CTIMP trial, which recruited between 03 Mar 2003 and 08 Feb 2012, formally ended on 31 May 2021.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Individual sites have statements of agreement that outline disclosure restrictions.